CLINICAL TRIAL: NCT02887248
Title: Phase II Study of Nanoparticle Albumin-bound Paclitaxel Plus Gemcitabine as First-line Therapy for the Treatment of Cisplatin-ineligible or Cisplatin-incurable Advanced Urothelial Carcinoma
Brief Title: Nab-paclitaxel Plus Gemcitabine as First-line Therapy for Cisplatin-ineligible or Cisplatin-incurable Advanced Urothelial Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrollment issues
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI GU 124
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Results first posted 2022-01-13 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2021-12

CONDITIONS: Urothelial Carcinoma; Bladder Cancer; Transitional Cell Carcinoma
Keywords: nab-paclitaxel; gemcitabine
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- nab-paclitaxel+gemcitabine (Experimental): Induction Phase: nab-paclitaxel (125 mg/m²) and gemcitabine (1000 mg/m²) by IV infusion on Days 1 and 8 of each 21-day cycle. Responding or stable patients will be treated with a minimum of 3 cycles and up to 6 cycles before starting the single agent maintenance therapy.
  Maintenance Phase: Patients completing 3-6 cycles of induction therapy with an objective response (complete or partial response) or stable disease will continue treatment with single agent nab-paclitaxel (260 mg/m²) by IV infusion every 21 days) until disease progression, intolerable toxicity or patient decision to discontinue treatment.
  Interventions: Drug: nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel — Induction: 125 mg/m² by intravenous (IV) infusion on Days 1 and 8 of each 21-day cycle for 3 to 6 cycles to be given with Gemcitabine.
  Maintenance: single agent nab-paclitaxel (260 mg/m²) by IV infusion every 21 days) until disease progression, intolerable toxicity or patient decision to discontinue treatment.
  Other Names: Abraxane
Drug: Gemcitabine — Induction: 1000 mg/m²) by IV infusion on Days 1 and 8 of each 21-day cycle for 3 to 6 cycles.
  Other Names: Gemzar

SUMMARY:
The purpose of this trial is to determine the benefit of the combination of nab-paclitaxel plus gemcitabine given for 6 cycles, followed by maintenance nab-paclitaxel alone, in patients with cisplatin-ineligible or cisplatin-incurable advanced urothelial carcinoma (UC).

DETAILED DESCRIPTION:
This open-label, non-randomized phase II trial evaluates the efficacy and toxicity of first-line treatment with a combination of gemcitabine and nab-paclitaxel, followed by maintenance therapy with nab-paclitaxel alone in patients with metastatic or locally advanced unresectable urothelial cancer. Two groups of patients are eligible: (1) patients who are poor candidates for treatment with cisplatin, and (2) patients with visceral metastases who are incurable and unlikely to derive long-term benefit from treatment with cisplatin-based regimens. Eligible patients will receive a minimum of 3 cycles and up to 6 cycles of treatment with the gemcitabine/nab-paclitaxel combination. Patients having an objective response or stable disease will continue maintenance treatment with single-agent nab-paclitaxel until disease progression, intolerable toxicity, or patient decision to discontinue treatment. Up to 55 patients are planned for enrollment.

ELIGIBILITY:
KEY POINTS:

Inclusion Criteria:

1. Histologically confirmed diagnosis of urothelial carcinoma (UC) that is either metastatic (any N+ M1) or locally advanced and unresectable (T4bN0). A component of urothelial (transitional cell) carcinoma is required.
2. Two groups of patients are eligible:

   1. Poor candidates for cisplatin-based chemotherapy based on the presence of ≥ 1 the following:

      * Glomerular filtration rate of 30-60 ml/min (Cockcroft-Gault formula)
      * ECOG performance status score of 2
      * Hearing loss (trouble communicating with hearing aids or hearing loss at ≤ 3 KHz)
      * Grade ≥3 heart failure
      * Age ≥80 years
      * Other concurrent illness which may make the patient a poor candidate for receiving cisplatin.

      Note: Enrollment of patients with 2 or more of these criteria should occur only after careful consideration by the treating physician regarding the patient's ability to tolerate combination chemotherapy.

      OR
   2. Poor prognosis and defined as cisplatin-incurable due to the presence of metastasis to at least one visceral site (these patients are not required to have any of the cisplatin-ineligibility criteria).

      * ECOG performance status score of 0, 1, or 2.
3. Measurable or evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
4. Patients with brain metastases are allowed if treatment was completed at least 4 weeks prior to study treatment, neurologic symptoms are minimal and stable during the preceding 4 weeks, and maintenance dexamethasone is not required.
5. Adequate hematologic, liver and kidney function.
6. Willingness and ability to comply with study requirements and give written informed consent.

Exclusion Criteria:

1. Previous systemic chemotherapy for UC with the exception of perioperative (neoadjuvant or adjuvant) treatment or treatment with concurrent chemoradiation for locally advanced disease. All of these treatments must have been completed more than 1 year previously.
2. Presence of small-cell or sarcomatoid component in tumor histology.
3. Women who are pregnant or breast-feeding.
4. Major surgical procedures ≤28 days of beginning study drug, or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
5. Cardiac diseases currently or within the last 6 months:
6. Inadequately controlled hypertension.
7. Currently receiving treatment with therapeutic doses of warfarin sodium. (A maximum daily dose of 1 mg will be permitted for port line patency. Low molecular weight heparin is allowed.)
8. Serious active infection at the time of treatment, or another serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
9. Known diagnosis of human immunodeficiency virus, hepatitis B or hepatitis C (screening for these diseases is not required.).
10. Presence of other active cancers, or history of treatment for invasive cancer ≤5 years previously. Patients with Stage I cancer who have received definitive local treatment and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (i.e., non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Hainsworth, MD, Study Chair — SCRI Development Innovations, LLC
Locations (5):
- United States (5):
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Florida Cancer Specialists-North, St. Petersburg, Florida
  - Florida Cancer Specialists-East, West Palm Beach, Florida
  - Tennessee Oncology, Nashville, Tennessee
  - Center for Cancer and Blood Disorders, Fort Worth, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nab-paclitaxel+Gemcitabine
Started | 3
Completed | 0
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: 6 Month Progression-free Survival (PFS6)
Description: The percentage of treated patients who are progression-free at 6 months after start of treatment, assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. Progressive disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest (nadir) sum since the treatment started, or the appearance of one or more new lesions. Requires not only 20% increase, but absolute increase of a minimum of 5 mm over sum.
Time Frame: up to 26 weeks
Population: Analysis was not done as the study ended early because of slow recruitment
Arm/Group | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Response Rate
Description: The proportion of patients with a confirmed complete or partial response (CR or PR) according to RECIST v1.1. CR = disappearance of all target lesions. PR = at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: every 3 cycles (9 weeks) until treatment discontinuation, an expected average of 1 year.
Population: Analysis was not done as the study ended early because of slow recruitment
Arm/Group | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 0

3. Secondary Outcome: Clinical Benefit Rate
Description: Defined as the proportion of patients with CR, PR, or stable disease (SD) according to RECIST v1.1. SD = neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest (nadir) sum of diameters since start of treatment.
Time Frame: every 3 cycles (9 weeks) until treatment discontinuation, an expected average of 1 year.
Population: Analysis was not done as the study ended early because of slow recruitment
Arm/Group | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Description: Defined as the time from Day 1 of study drug administration to disease progression or death on study.
Time Frame: every 9 weeks until disease progression or death on study, an expected average of 1 year. Patients with progressive disease will be followed every 3 months for the first year and every 6 months thereafter up to 5 years.
Population: Analysis was not done as the study ended early because of slow recruitment
Arm/Group | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 0

5. Secondary Outcome: The Number of Participants With Grade 3/4/5 Adverse Events (AEs) as a Measure of Safety.
Description: The reported incidence of AEs with an onset on or after the initiation of therapy will be graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-paclitaxel+Gemcitabine
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 year
Arm/Group | Nab-paclitaxel+Gemcitabine
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel+Gemcitabine (N=3)
Hypotension (Vascular disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nab-paclitaxel+Gemcitabine (N=3)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (5)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Asthenia (General disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (8)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 2 (4)
Gout (Metabolism and nutrition disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (4)
Hypotension (Vascular disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (3)
Malaise (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Oedema (General disorders) | 1 (3)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT02887248/Prot_SAP_000.pdf